CLINICAL TRIAL: NCT05160324
Title: T1-T2 Breast Cancer: Comparison Between Removal and Preservation of Axillary Lymph Nodes in the Presence of Sentinel Lymph Node Metastases (SINODAR ONE)
Brief Title: T1-T2 Breast Cancer: Comparison Between Removal and Preservation of Axillary Lymph Nodes (SINODAR ONE)
Acronym: SINODAR ONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Humanitas per la Ricerca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1317
Record Dates: First submitted 2021-11-19; First posted 2021-12-16 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer
Keywords: axillary dissection, axillary lymph preservation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Axillary dissection (standard treatment) (Active Comparator): Axillary dissection in women with sentinel lymph node metastases.
  (removal of at least 10 lymph nodes recommended)
  Interventions: Procedure: Removal of axillary lymph nodes.
- Preservation of axillary lymph nodes (Experimental): Omission of Axillary dissection in women with sentinel lymph node metastases.
  Interventions: Procedure: Preservation of axillary lymph nodes

INTERVENTIONS:
Procedure: Removal of axillary lymph nodes. — Axillary dissection in patients with positive sentinel lymph node
  Arms: Axillary dissection (standard treatment)
Procedure: Preservation of axillary lymph nodes — Preservation of axillary lymph nodes in patients with positive sentinel lymph node
  Arms: Preservation of axillary lymph nodes

SUMMARY:
Italian Multicentric non inferiority two-arm randomized clinical trial to verify that the experimental treatment (omission of axillary lymph node intervention) in the presence of sentinel lymph node metastases does not lead to a significant worsening in survival or in the risk of locoregional recurrence compared to standard treatment (removal of I-II level of axillary lymph nodes).

DETAILED DESCRIPTION:
Detailed Description:

The trial is a non-inferiority trial; patients, depending on intra-operative or post-operative sentinel lymph node assessment, are randomly assigned to one of the two intervention groups:

group 1: removal of I-II level of axillary lymph nodes (standard treatment). Removal of at least 10 lymph nodes is recommended.

group 2: no axillary lymph nodes dissection (experimental treatment). Patients for whom sentinel lymph node cannot be found, will undergo complete dissection of the axillary cavity as required by international guidelines.

After surgery, according to their bio-pathological profile and to the international guidelines criteria, patients will be able to receive:

* no further treatment
* complementary radiotherapy
* adjuvant medical therapy (chemo and / or hormone therapy).

Patients will be checked for at least 5 years in the following ways:

* six-monthly clinical examination for the first 5 years and yearly thereafter
* mammography + annual breast ultrasound
* annual axillary ultrasound in cases not subjected to dissection.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 ≤75 years old
* Breast cancer with infiltrating histology
* Tumor size ≤50 mm (T1 - T2)
* Clinically and ultrasound node-negative (cN0) breast cancer
* No distant metastases (M0)
* No neoadjuvant therapy
* Negative history of previous infiltrating neoplasm
* Maximum number of metastatic sentinel lymph nodes: 2
* Lymph node macro-metastases > 2mm

Exclusion Criteria:

* Pregnancy or breastfeeding in progress
* Inflammatory breast cancer
* Breast cancer in situ
* Synchronous contralateral breast cancer
* Co-morbidities such as to preclude the possible use of adjuvant therapy
* Conditions that make it impossible to carry out a regular follow-up
* Other malignancies within the previous 3 years (except carcinoma in situ of the uterine cervix, basalioma or squamous cell ca or non-melanoma skin ca)
* Breast cancer with non-infiltrating or inflammatory histotype
* Tumor size> 50 mm
* No sentinel lymph nodes identified
* No positive sentinel lymph nodes (pN0)
* Positive sentinel lymph node number > 2
* Lymph node micro-metastases <= 2

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 889 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5 years of follow up after surgery
  Evaluating whether, in women operated for breast cancer (T1-T2) with sentinel lymph node metastases, axillary lymph node conservation is associated with a clinically relevant prognostic worsening (OS). For all the Outcomes Statistical analysis included Kaplan-Meier Product Limit Estimator and the log-rank test

SECONDARY OUTCOMES:
Regional Disease Free Survival (RDFS) | 5 years of follow up after surgery
  Evaluating whether axillary lymph node preservation is associated with a clinically relevant increase of local recurrence rate (ipsilateral axillary and supraclavicular lymph nodes).
Disease-free distance survival (DDFS) | 5 years of follow up after surgery
  Evaluating whether axillary lymph node preservation is associated with a clinically relevant increase in distant recurrence rate.

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Tinterri, MD, Principal Investigator — Istituto Clinico Humanitas

REFERENCES:
- [Derived] Tinterri C, Canavese G, Gatzemeier W, Barbieri E, Bottini A, Sagona A, Caraceni G, Testori A, Di Maria Grimaldi S, Dani C, Boni L, Bruzzi P, Fernandes B, Scorsetti M, Zambelli A, Gentile D; SINODAR-ONE Collaborative Group. Sentinel lymph node biopsy versus axillary lymph node dissection in breast cancer patients undergoing mastectomy with one to two metastatic sentinel lymph nodes: sub-analysis of the SINODAR-ONE multicentre randomized clinical trial and reopening of enrolment. Br J Surg. 2023 Aug 11;110(9):1143-1152. doi: 10.1093/bjs/znad215. PMID 37471574